CLINICAL TRIAL: NCT01554319
Title: Phase-I Study in Healthy Male Subjects to Investigate Safety, Tolerability and Pharmacokinetics of Orally Inhaled Multiple Doses of SB010, a Human GATA-3-specific DNAzyme Solution for Nebulisation
Brief Title: Safety, Tolerability, and Pharmacokinetics After Multiple Doses of Orally Inhaled DNAzyme Solution for Nebulisation in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sterna Biologicals GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB010/02/2011; 2011-005782-20 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-14 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Antisense oligonucleotide; Asthma; Healthy subjects; Phase 1; Transcription factor GATA-3; Oral inhalation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB010 (Experimental): The drug will be administered in phosphate-buffered saline solution, inhaled over 5 - 10 min, using a hand-held inhalation device.
  Initial single dose on Day 1 (single-dose PK profile); after 48 h washout, twice-daily with a dosing interval of 12 h for 9 consecutive days (Days 3 to 11); last inhalation on Day 12.
  Interventions: Drug: SB010
- Placebo (Placebo Comparator): The placebo (phosphate-buffered saline) is administered as a solution, inhaled over 5 - 10 min, using a hand-held inhalation device.
  Initial single dose on Day 1 (single-dose PK profile); after 48 h washout, twice-daily with a dosing interval of 12 h for 9 consecutive days (Days 3 to 11); last inhalation on Day 12.
  Interventions: Drug: Placebo (phosphate-buffered saline)

INTERVENTIONS:
Drug: SB010 — Three ascending dose groups are planned (Groups A, B, C), each consisting of 12 male subjects. Each of the 3 dose groups will be divided into 2 subgroups. First subgroup: 4 subjects (n=3 active compound, n=1 placebo); second subgroup: 8 subjects (n=6 active compound, n=2 placebo).
  Each dose group will be investigated with a new group of 12 subjects (n=9 active compound, n=3 placebo). Dose escalation to next dose level will occur after satisfactory review of safety and tolerability and after review of the pharmacokinetic data (exposure control) of the preceding dose cohorts by the Safety Board.
  Dose group A : 5 mg hgd40/2 mL; Dose group B: 10 mg hgd40/2 mL; Dose group C: 20 mg hgd40/2 mL.
  Arms: SB010
Drug: Placebo (phosphate-buffered saline) — Three ascending dose groups are planned (Groups A, B, C), each consisting of 12 male subjects. Each of the 3 dose groups will be divided into 2 subgroups. First subgroup: 4 subjects (n=3 active compound, n=1 placebo); second subgroup: 8 subjects (n=6 active compound, n=2 placebo).
  Each dose group will be investigated with a new group of 12 subjects (n=9 active compound, n=3 placebo). Dose escalation to next dose level will occur after satisfactory review of safety and tolerability and after review of the pharmacokinetic data (exposure control) of the preceding dose cohorts by the Safety Board.
  Arms: Placebo

SUMMARY:
Asthma is a chronic inflammatory bronchial disorder with three distinct components: airway hyper-responsiveness (respiratory hypersensitivity), airway inflammation, and intermittent airway obstruction. One of the characteristics of the disease is an inflammatory reaction of the immune system caused by cytokine production. A substantial number of asthma patients do not satisfactorily respond to steroid therapy and consequently have an unmet medical need for novel targeted therapies with improved specificity, tolerability, and compliance.

Novel therapeutic strategies for the treatment of chronic inflammatory diseases by targeting early disease-causing mechanisms are a promising approach for the treatment of asthma. The transcription factor GATA-3 plays a key role in mediating the asthmatic immune response and has been shown to be necessary and sufficient for the production of cytokines interleukin (IL)-4, IL-5, and IL-13. The active principle hgd40 of the investigational medicinal product SB010 belongs to a new class of antisense oligonucleotide therapeutics, the 10-23 DNA (deoxyribonucleic acid)zymes (antisense oligonucleotide). DNAzymes are catalytically active nucleic acids that cleave complementary RNA (ribonucleic acid) molecules. By cleaving GATA-3 mRNA, hgd40 reduces specific cytokine production and thereby reduces key features of allergic airway inflammation.

DNAzymes are generated completely by chemical synthesis and can be produced under Good Manufacturing Practice (GMP) controlled conditions. The DNAzymes are not biological drugs, i.e. they are not generated by use of any living organism including cell culture or bacteria. The molecules are highly water-soluble and will be applied as solution directly in their synthesized form.

The current study will evaluate the safety and tolerability of increasing multiple doses of inhaled SB010 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been informed both verbally and in writing about the objectives of the clinical trial, the methods, the anticipated benefits and potential risks and the discomfort to which he may be exposed, and has given written consent to participation in the trial prior to trial start and any trial-related procedure.
* Healthy male Caucasian subject, aged between 18 and 45 years (inclusive), assessed as healthy based on a screening examination including medical history without clinically relevant pathologies, physical examination, vital signs, ECG assessment, pulmonary function testing, and clinical laboratory results.
* Body weight according to a body mass index ≥18.0 and ≤29.0 kg/m2, and a body weight ≥60 and ≤90 kg.
* Non-smokers or ex-smokers who had stopped smoking for at least 5 years prior to start of the clinical study.
* Ability to inhale in an appropriate manner (Subjects will be trained to inhale using the AKITA2 APIXNEB® device with a placebo medication at the screening visit).
* The subject must agree:

  * to use two methods of contraception in combination with his female partner, if she is of childbearing potential; this combination of contraceptive methods must be used from screening until at least 6 months after the last dose of IMP. At least one of the contraception methods must be a barrier contraception method. Contraceptive methods allowed include the following: condoms, diaphragm in combination with a spermicide, intrauterine device as well as for female partners oral contraception, contraception implants, OR
  * not to be sexually active at screening and accept using double-barrier contraception should he become sexually active during or within 6 months after the last dose of IMP, OR
  * to have been surgically sterilised prior to screening and accept to use a barrier method of contraception as well, OR
  * to have a partner who is post-menopausal and has had her last natural menstruation at least 24 months prior to screening, OR
  * to have a partner who has had a hysterectomy prior to screening, OR
  * to have a partner who has been surgically sterilised prior to screening

All assessments will be performed within 2 to 14 days prior to first dose with the active compound or placebo.

Exclusion Criteria:

* History or current evidence of clinically relevant allergies or idiosyncrasy to any drug or food.
* History of allergic reactions to any active or inactive component of the study medication.
* Any history of allergic rhinitis or atopic disease. Subjects with total immunoglobulin E levels >150 kU/L will be excluded.
* History or current evidence of any clinically relevant pulmonary, cardiovascular, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological, or psychiatric disease within the last 2 years.
* ECG abnormalities of clinical relevance (e.g., QTc according to Bazett's ≥440 ms, PR ≥210 ms; or QRS ≥120 ms).
* Subjects with a resting heart rate between 50 bpm and 90 bpm (inclusive), systolic blood pressure between 100 mmHg and 140 mmHg (inclusive), diastolic blood pressure between 60 mmHg and 90 mmHg (inclusive).
* Proneness to orthostatic dysregulation, fainting, or blackouts.
* History or presence of any malignancy except for basalioma.
* Abnormalities in clinical chemical or haematological variables considered medically relevant by the investigator. Values for total leukocytes and neutrophils, gamma-glutamyltranspeptidase, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, lactate dehydrogenase, bilirubin, and serum creatinine should be within normal ranges.
* Chronic or acute infections.
* Positive results in any of the following virology tests: human immunodeficiency virus antibodies and antigen, Anti-hepatitis B-core antibody, hepatitis B surface antigen and anti-hepatitis C virus antibody.
* Positive drug screen.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Limiting dose of inhaled ascending multiple doses of SB010. | Up to Day 71±4 (maximum 89 days for a particular patient)
  Safety will be monitored as adverse events, vital signs, clinical chemistry, haematology, coagulation, urinalysis, electrocardiogram, pulmonary function testing, body temperature, overall tolerability.

SECONDARY OUTCOMES:
Number of participants with any dose-limiting adverse effects, after multiple doses of inhaled SB010. | Screening examination (Day 14 to 2 before first drug administration); Study period (Day 1 to 15); Follow-up visit (Days 23±2); Follow-up phone call (Day 41±3); End-of-study visit (Day 71±4). Maximum of 89 days for a particular subject.
  Safety will be monitored as adverse events, vital signs, clinical chemistry, haematology, coagulation, urinalysis, electrocardiogram, pulmonary function testing, body temperature, overall tolerability.
Plasma concentration of hgd40 over time after multiple inhaled doses of SB010. | Study period (Day 1 to 15).
  The following pharmacokinetic parameters will be determined over 15 days using plasma samples, after a single dose on Day 1 and after repeated dosing at steady state on Day 12:
  Area under the plasma concentration-time curve: from 0 to 12h, over 12h (dosing interval) after the last administration in steady state, and extrapolated to infinity.
  Concentration maximum.
  Time of maximum concentration.
  Terminal disposition rate constant and the respective half-life.
  Accumulation index.
Plasma concentration of hgd40 over time after multiple inhaled doses of SB010 (Dose proportionality over time). | Study period (Day 1 to 15).
  Dose proportionality# after a single dose on Day 1 and after repeated dosing at steady state on Day 12 will be assessed across doses using the power model.
  #Dose proportionality implies linear pharmacokinetics. The rates of absorption, distribution, metabolism, and elimination remain constant over the dose range. Thus, plasma concentration, area under the plasma concentration-time curve, maximum plasma concentration, and urinary recovery should increase in direct proportion to the dose.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Timmer, MD, Principal Investigator — CRS-Mannheim GmbH, Germany
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany